CLINICAL TRIAL: NCT03893708
Title: The Power of Yoga: Investigating the Feasibility and Preliminary Effects of Yoga on Excessive Gestational Weight Gain
Brief Title: Investigating the Feasibility and Preliminary Effects of Yoga on Excessive Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Kripalu Center for Yoga and Health (Other)
Responsible Party: Principal Investigator, Jennifer Huberty, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007808; FP00012624 (Other Grant/Funding Number: Kripalu Center for Yoga and Health)
Record Dates: First submitted 2019-03-19; First posted 2019-03-28 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Weight Gain
Keywords: pregnancy; prenatal yoga; excessive gestational weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal yoga (Experimental): Each class will be outlined as follows: 1) opening greeting/intention setting, 2) pranayama (i.e., breathing exercises), 3) warm-up/sun salutations (i.e., flowing sequence), 4) yoga sequence (e.g., combination of sun salutations, vinyasa, and standing, seated, and/or balancing poses), 5) cool-down 6) Savasana (i.e., final resting pose), and 7) class closing. Meditation and breath awareness (e.g., linking each movement with breath) will be emphasized throughout each class. All classes will focus on safety and alignment and be appropriate for women during pregnancy by incorporating modifications to poses/exercises as necessary (e.g., yoga block, strap). Certified yoga instructors with a bachelors degree in a health related field and experience teaching pregnant women will instruct all yoga classes. Participants will be provided with a 'yoga during pregnancy' safety packet that includes a list of prenatal yoga poses that women may do at their own leisure at home.
  Interventions: Behavioral: Prenatal yoga
- Pregnancy education (Active Comparator): Participants will be asked to attend a group-based pregnancy education group (similar to a birth education class). The class format will include a didactic portion followed by group discussion (N=12). The following evidence-based topics (based on the American College of Obstetrics and Gynecologists) to be discussed may include (but not limited to): financial management in preparation for baby, preparing for labor and delivery, transitioning into motherhood, sleep hygiene, and baby bonding. A labor and delivery nurse and certified Dula will instruct all classes.
  Interventions: Behavioral: Pregnancy education

INTERVENTIONS:
Behavioral: Prenatal yoga — The prenatal yoga classes will be offered at Urban Wellness (2024 N. 7th St., Phoenix, AZ 85006). Classes will be offered Tuesdays's from 4:15-5:30 pm and Saturday's from 9:00-10:15 am. Participants will be able to attend both classes if they so choose but are only asked to attend 1/week. Participants will be asked to arrive to class at least 10 minutes early in order for the research team to collect their weight in a private room. Additionally, if participants have attended at least 70% of classes (1 per week for 8/12 weeks), participants will be able to attend sessions up until birth (beyond the 12-week intervention) if they so choose. If participants decide to attend classes beyond the 12-week intervention the investigators will continue to collect their weight at each session.
  Arms: Prenatal yoga
Behavioral: Pregnancy education — Pregnancy education classes will be offered at the Arizona Biomedical Collaborative Building on ASU Phoenix Campus. Classes will be offered on Tuesday's from 5:30-6:45 pm and Saturday's from 9:00-10:15 am. Participants will be able to attend both classes if they so choose but are only asked to attend 1/week. Participants will be asked to arrive to class at least 10 minutes early in order for the research team to collect their weight in a private room. Additionally, if participants have attended at least 70% of classes (1 per week for 8/12 weeks), participants will be able to attend sessions up until birth (beyond the 12-week intervention) if they so choose. If participants decide to attend classes beyond the 12-week intervention the investigators will continue to collect their weight at each session.
  Arms: Pregnancy education

SUMMARY:
This study will test the feasibility (i.e., acceptability, demand) of a 12-week prenatal yoga intervention on excessive gestational weight gain (GWG) in pregnant women in the second trimester (enrolled at 12-24 weeks). Participants will be randomized into the prenatal yoga intervention or a pregnancy education (e.g., information on preparing for motherhood, labor and delivery etc.) control group. Participants in both groups will be asked to attend one 75 minute class per week.

The investigators hypothesize that prenatal yoga intervention will be feasible for pregnant women.

The study aims are as follows:

Primary Aim: Determine the feasibility (i.e., acceptability, demand) of a 12-week prenatal yoga intervention in pregnant women. In a randomized controlled pilot study comparing prenatal yoga to a pregnancy education control condition, the investigators will assess 1) acceptability (defined as satisfaction, intent to continue use, perceived appropriateness) and 2) demand (defined as attendance/adherence).

Exploratory Aim 1: Ascertain the preliminary effects of prenatal yoga on excessive GWG [i.e., weight gain exceeding Institute of Medicine (IOM) recommendations]. The investigators will compare weight change between intervention and control groups.

Exploratory Aim 2: Explore the potential mediators (i.e., mindfulness, self-regulation) on the effect of prenatal yoga on excessive GWG.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-46 years of age (childbearing age)
* Primiparous (women giving birth for the first time)
* 12-24 weeks gestation at onset of intervention
* Reside in the Phoenix Metropolitan area
* Singleton pregnancy
* English speaking
* Not planning on moving before giving birth
* Can attend at least one session per week

Exclusion Criteria:

* Current alcohol or substance abuse
* Engage in ≥150 min of physical activity
* Participation in ≥30 minutes/week of yoga or contemplative practice (i.e., meditation, qigong) for the previous six months
* Pre-pregnancy BMI ≥40 or <18.5
* Denial of physical activity participation from a physician (PARmed-X for pregnancy)

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability via satisfaction survey at post-intervention | post-intervention (12-weeks)
  Acceptability (defined as satisfaction, intent to continue use, perceived appropriateness); Benchmarks for acceptability include ≥70% of the sample will report the yoga intervention to be a satisfactory, useful, and appropriate modality to prevent excessive GWG.
Demand (attendance/adherence) of yoga intervention | Weekly (during 12-week intervention)
  Demand was measured using attendance/adherence to the yoga intervention. Attendance was tracked by a researcher who was present at each yoga session. Benchmarks for demand include ≥60% of participants in each group will attend one class per week.

SECONDARY OUTCOMES:
Number of participants with excessive GWG (total GWG from baseline to delivery) | Weekly (during 12-week intervention) and at delivery (up to 42 weeks gestation)
  Weight gain exceeding IOM recommendations
Mindfulness (mean change from baseline) | Baseline, post-intervention (12-weeks)
  Self-report mindfulness scores via Mindful Attention Awareness Scale (MAAS); 15-item questionnaire with score ranges 1-6. Higher scores reflect higher levels of dispositional mindfulness.
Self-awareness (mean change from baseline) | Baseline, post-intervention (12-weeks)
  Self-report self-awareness scores via Self-Awareness Outcomes Questionnaire (SAOQ); Consists of 38 items measuring 4 subscales (reflective self-development, acceptance, proactive at work, and emotional costs). Score ranges for each subscale are between 1-5. Higher scores represent a greater frequency of experienced outcomes.
Emotion Regulation (mean change from baseline) | Baseline, post-intervention (12-weeks)
  Self-report emotion regulation scores via Emotional Regulation Questionnaire (ERQ); Consists of 10 items measuring 2 subscales (reappraisal items, suppression items). Score ranges for each subscale are between 1-7. The higher the scores, the greater the use of the emotional regulation strategy.
Sleep Quality (mean change from baseline) | Baseline, post-intervention (12-weeks)
  Self-report sleep quality via Pittsburgh Sleep Quality Index (PSQI); Consists of 10-items. In scoring the PSQI, seven component scores are derived ranging from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PHD, Principal Investigator — Arizona State University
Locations (2):
- United States (2):
  - Arizona Biomedical Collaborative (ASU), Phoenix, Arizona
  - Urban Wellness, Phoenix, Arizona

IPD SHARING:
Plan to Share IPD: No
Consent forms indicate that data will not be shared with anyone other than those listed on the study team.